CLINICAL TRIAL: NCT02464280
Title: Validation of Tomosynthesis for Indications for Clinical Questions Concerning Pathologies of the Chest and Skeletal Structures: When Can CT Been Omitted?
Brief Title: Tomosynthesis of Pathologies of the Chest and Skeletal Structures in Comparison to CT
Status: Terminated | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SNCTP000001072
Record Dates: First submitted 2014-09-25; First posted 2015-06-08 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lung Disease; Wrist Fracture
Keywords: Tomosynthesis; osteosynthetic implant; CT; monitoring
MeSH Terms: conditions — Lung Diseases; Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients scheduled for lung imaging: Patients with lung changes and scheduled for lung imaging will undergo:
  * the scheduled conventional X-ray examination
  * the scheduled CT scan
  * the tomosynthesis scan
  Interventions: Other: Tomosythesis scan of the lung or the wrist; Other: CT scan of the lung or the wrist; Other: conventional X-ray of the lung or the wrist
- Patients scheduled for wrist imaging: Patients with wrist fracture or with osteoprotetic material in the wrist and scheduled for wrist imaging will undergo:
  * the scheduled conventional X-ray examination
  * the scheduled CT scan
  * the tomosynthesis scan
  Interventions: Other: Tomosythesis scan of the lung or the wrist; Other: CT scan of the lung or the wrist; Other: conventional X-ray of the lung or the wrist

INTERVENTIONS:
Other: Tomosythesis scan of the lung or the wrist — All study participants will undergo Tomosynthesis imaging of the lung or the wrist. The radiation dose of each method will be recorded.
Other: CT scan of the lung or the wrist — All study participants will undergo CT imaging of the lung or the wrist, for which they where originally scheduled. The radiation dose of each method will be recorded.
Other: conventional X-ray of the lung or the wrist — All study participants will undergo conventional X-ray of the lung or the wrist, for which they where originally scheduled. The radiation dose of each method will be recorded.

SUMMARY:
The investigators propose tomosynthesis as a imaging method in between of x-ray and CT. The expected value of this project is the definition of proven indications for tomosynthesis, which allow replacing CT. Specific goals are the early detection of pulmonary consolidations / parenchymal changes as well as the monitoring of patients with ostesynthetic implants.

DETAILED DESCRIPTION:
The investigators propose tomosynthesis as a imaging method in between of x-ray and CT. The expected value of this project is the definition of proven indications for tomosynthesis, which allow replacing CT. Specific goals are the early detection of pulmonary consolidations / parenchymal changes as well as the monitoring of patients with ostesynthetic implants.

This is a prospective, single-center, non-randomised, non-blinded trial with Tomosyntheis of Patients referred to the investigators institution to assess lung alterations and bone structure. All patients will undergo chest x-ray and tomosynthesis after informed consent. In addition they will undergo an ultralow-dose CT, wich is used as standart reference. The radiation dose of each method will be recorded. After completion of these three examinations, the participation in the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for evaluation of lung-changes
* Patients scheduled for evaluation of the wrist after fracture or surgery

Exclusion Criteria:

* general contraindications for x-Ray
* general contraindications for CT
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population included in this study are patients who are referred to our hospital for evaluation of lung-changes or evaluation of the wrist after fracture or surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Non-Inferiority CT | when scheduled for x-ray - 52 weeks
  Value of Tomosynthesis-image information compared to CT

SECONDARY OUTCOMES:
Superiority to x-ray | when scheduled for x-ray - 52 weeks
  Value of Tomosynthesis-image information compared to x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Thoams Frauenfelder, MD, Principal Investigator — University Hospital Zurich, Radiology
Locations (1):
- University Hospital Zurich - Diagnostic Radiology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No